CLINICAL TRIAL: NCT04250363
Title: A Phase Ib, Randomized, Double-Blind, Placebo Controlled, Sequential Study of Single Oral Doses of M5717 to Explore the Chemoprophylactic Activity of M5717 in a Controlled PISPZ Challenge Model in Healthy Participants
Brief Title: Chemoprophylactic Activity of M5717 in PfSPZ Challenge Model
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: MS201618_0003; 2019-003414-14 (EudraCT Number); 203481/Z/16/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2023-11

CONDITIONS: Healthy
Keywords: Healthy Participants; M5717; Malaria; Plasmodium falciparum
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Early liver stage: Pooled Placebo (Placebo Comparator): Participants received single dose of placebo matched to M5717 capsule on Day 1 after 2 hours of Plasmodium falciparum Sporozoite (PfSPZ) (3200 sporozoites per injection) intravenous (IV) inoculation administration on Day 1.
  Interventions: Biological: PfSPZ Challenge; Drug: Palcebo
- Early liver stage: 30 mg M5717 (Experimental): Participants received single dose of M5717 30 mg capsule on Day 1 after 2 hours of PfSPZ (3200 sporozoites per injection) IV inoculation administration on Day 1.
  Interventions: Biological: PfSPZ Challenge; Drug: M5717 30 mg
- Early liver stage: 60 mg M5717 (Experimental): Participants received single dose of M5717 60 mg capsule on Day 1 after 2 hours of PfSPZ (3200 sporozoites per injection) IV inoculation administration on Day 1.
  Interventions: Biological: PfSPZ Challenge; Drug: M5717 60 mg
- Early liver stage: 80 mg M5717 (Experimental): Participants received single dose of M5717 80 mg capsule on Day 1 after 2 hours of PfSPZ (3200 sporozoites per injection) IV inoculation administration on Day 1.
  Interventions: Biological: PfSPZ Challenge; Drug: M5717 80 mg
- Early liver stage: 100 mg M5717 (Experimental): Participants received single dose of M5717 100 mg capsule on Day 1 after 2 hours of PfSPZ (3200 sporozoites per injection) IV inoculation administration on Day 1.
  Interventions: Biological: PfSPZ Challenge; Drug: M5717 100 mg
- Early liver stage: 200 mg M5717 (Experimental): Participants received single dose of M5717 200 mg capsule on Day 1 after 2 hours of PfSPZ (3200 sporozoites per injection) IV inoculation administration on Day 1.
  Interventions: Biological: PfSPZ Challenge; Drug: M5717 200 mg
- Late liver stage: Pooled Placebo (Experimental): Participants received single dose of placebo matched to M5717 capsule on Day 5 after 96 hours of PfSPZ (3200 sporozoites per injection) IV inoculation administration on Day 1.
  Interventions: Biological: PfSPZ Challenge; Drug: Placebo
- Late liver stage: 60 mg M5717 (Experimental): Participants received single dose of M5717 60 mg capsule on Day 5 after 96 hours of PfSPZ (3200 sporozoites per injection) IV inoculation administration on Day 1.
  Interventions: Biological: PfSPZ Challenge; Drug: M5717 60 mg
- Late liver stage: 100 mg M5717 (Experimental): Participants received single dose of M5717 100 mg capsule on Day 5 after 96 hours of PfSPZ (3200 sporozoites per injection) IV inoculation administration on Day 1.
  Interventions: Biological: PfSPZ Challenge; Drug: M5717 100 mg
- Late liver stage: 200 mg M5717 (Experimental): Participants received single dose of M5717 200 mg capsule on Day 5 after 96 hours of PfSPZ (3200 sporozoites per injection) IV inoculation administration on Day 1.
  Interventions: Biological: PfSPZ Challenge; Drug: M5717 200 mg

INTERVENTIONS:
Biological: PfSPZ Challenge — Participants received 3200 units of Plasmodium falciparum sporozoites by DVI on Day 1.
Drug: Palcebo — Participants received single oral dose of placebo matched to M5717 capsule on Day 1.
  Arms: Early liver stage: Pooled Placebo
Drug: M5717 30 mg — Participants received 30 mg single oral dose of M5717 capsule on Day 1.
  Arms: Early liver stage: 30 mg M5717
Drug: M5717 60 mg — Participants received 60 mg single oral dose of M5717 capsule on Day 1.
  Arms: Early liver stage: 60 mg M5717
Drug: M5717 80 mg — Participants received 80 mg single oral dose of M5717 capsule on Day 1.
  Arms: Early liver stage: 80 mg M5717
Drug: M5717 100 mg — Participants received 100 mg single oral dose of M5717 capsule on Day 1.
  Arms: Early liver stage: 100 mg M5717
Drug: M5717 200 mg — Participants received 200 mg single oral dose of M5717 capsule on Day 1.
  Arms: Early liver stage: 200 mg M5717
Drug: Placebo — Participants received single oral dose of placebo matched to M5717 capsule on Day 5.
  Arms: Late liver stage: Pooled Placebo
Drug: M5717 60 mg — Participants received 60 mg single oral dose of M5717 capsule on Day 5.
  Arms: Late liver stage: 60 mg M5717
Drug: M5717 100 mg — Participants received 100 mg single oral dose of M5717 capsule on Day 5.
  Arms: Late liver stage: 100 mg M5717
Drug: M5717 200 mg — Participants received 200 mg single oral dose of M5717 capsule on Day 5.
  Arms: Late liver stage: 200 mg M5717

SUMMARY:
The main purpose of this study was to assess the chemoprophylactic activity and dose-exposure-response relationship of single oral dose of M5717 administered after direct intravenous inoculation (DVI) of Plasmodium falciparum sporozoite (PfSPZ) challenge in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation, including no clinically significant abnormality identified on physical examination or laboratory evaluation and no active clinically significant disorder, condition, infection or disease that would pose a risk to participant safety or interfere with the study evaluation, procedures or completion
* Participants who have a body weight within 50 to 100 kilograms (kg) and body mass index within the range 19.0 to 29.9 kilograms per meter square (kg/m2) (inclusive)
* Male participants, during the study intervention period and for at least 120 days after the day of the study intervention dose (covering a full sperm cycle of 90 days starting after 5 half lives of last dose of study intervention: - refrain from donating sperm plus, either - abstain from intercourse with a woman of childbearing potential (WOCBP) or - use a male condom, when having sexual intercourse with a WOCBP, who is not currently pregnant, and advise her to use a highly effective contraceptive method with a failure rate of less than (<) 1 percent (%) per year, since a condom may break or leak
* Female participants who are: - not a WOCBP; - at least 1 year post-menopausal (amenorrhea greater than or equal to [>=] 12 months and follicle-stimulating hormone [FSH] >= 40 milli-international units per milliliter [mIU/mL]) at screening; - surgically sterile (bilateral oophorectomy, hysterectomy or bilateral salpingectomy; tubal ligation alone is not sufficient)
* Participants who are capable of giving signed informed consent, which includes compliance with the requirements (including mandatory intake of rescue medication to participants who have been administered the investigational Plasmodium falciparum sporozoite challenge) and restrictions listed in the informed consent form (ICF) and this protocol
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants with 12-Lead electrocardiogram (ECG) outside normal range (QTcF greater than [>] 450 milli seconds [ms], pulse rate [PR] > 215 ms, or QRS > 120 ms) and deemed clinically relevant by the Investigator
* Supine systolic blood pressure > 140 or < 90 millimeter of mercury (mmHg), diastolic blood pressure > 90 or < 50 mmHg, and pulse rate > 90 or < 50 beats per minute (min) at screening and at admission on Day -1 (any abnormal blood pressure or pulse rate results may be repeated once and if the repeat result is within the normal range, it is not considered to have met the exclusion criterion)
* Seropositive for human immunodeficiency virus (HIV) I and II antibody or antigen), hepatitis B virus (HBV; hepatitis B surface antigen [HBsAg]), or hepatitis C virus (HCV; antibody) tests
* Liver function tests above the upper limit of normal (ULN) (> 3 x ULN) the day before DVI / study intervention administration (Day -1)
* History or presence of diagnosed food or known drug allergies (including but not limited to allergy to any of the antimalarial rescue medications to be used in the study), or history of anaphylaxis or other severe allergic reactions
* Participant with a whole blood donation or loss of > 450 mL within 60 days before administration of study drug or unwilling to defer blood donations for 6 months
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- [Derived] van der Plas JL, Kuiper VP, Bagchus WM, Bodding M, Yalkinoglu O, Tappert A, Seitzinger A, Spangenberg T, Bezuidenhout D, Wilkins J, Oeuvray C, Dhingra SK, Thathy V, Fidock DA, Smidt LCA, Roozen GVT, Koopman JPR, Lamers OAC, Sijtsma J, van Schuijlenburg R, Wessels E, Meij P, Kamerling IMC, Roestenberg M, Khandelwal A. Causal chemoprophylactic activity of cabamiquine against Plasmodium falciparum in a controlled human malaria infection: a randomised, double-blind, placebo-controlled study in the Netherlands. Lancet Infect Dis. 2023 Oct;23(10):1164-1174. doi: 10.1016/S1473-3099(23)00212-8. Epub 2023 Jul 3. PMID 37414066
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS201618_0003
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 39 participants (27 participants in early liver stage group and 12 participants in late liver stage group) were enrolled and randomized for treatment at single site in Netherlands.
Period: Overall Study
Arm/Group | Early Liver Stage: Pooled Placebo | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717 | Late Liver Stage: Pooled Placebo | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
Started | 6 | 3 | 6 | 6 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 6 | 3 | 6 | 6 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis population (SAF) included all intent to treat (ITT) participants, who have been inoculated using a Direct Intravenous Inoculation (DVI) of PfSPZ and who were administered one dose of study intervention (M5717 or placebo). ITT population included all participants, who were randomized to study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Liver Stage: Pooled Placebo | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717 | Late Liver Stage: Pooled Placebo | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717 | Total
Number analyzed (Participants) | 6 | 3 | 6 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 6 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 39
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 3 | 0 | 0 | 2 | 1 | 2 | 1 | 11
  Male | 6 | 3 | 4 | 3 | 3 | 3 | 1 | 2 | 1 | 2 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 3 | 5 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 38
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
  White | 5 | 3 | 6 | 5 | 3 | 2 | 3 | 2 | 3 | 3 | 35
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Early Liver Stage: Number of Participants Over Time With Positive Parasitemia
Description: Number of participants with positive parasitemia defined as first positive quantitative polymerase chain reaction (qPCR) outcome equal or greater than 100 asexual parasites per milliliter (mL) of blood within 28 days of PfSPZ challenge.
Time Frame: Early Liver Stage: From Day 1 up to Day 28
Population: Per-protocol (PP) analysis set included all SAF participants who comply with the protocol and meet no criteria that could impact the proper evaluation of key objectives of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Liver Stage: Pooled Placebo | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717
Number analyzed (Participants) | 6 | 3 | 6 | 6 | 3 | 3
Participants | 6 | 3 | 2 | 1 | 0 | 0

2. Primary Outcome: Late Liver Stage: Number of Participants Over Time With Positive Parasitemia
Description: as for outcome 1
Time Frame: Late Liver Stage: From Day 5 up to Day 32
Population: PP analysis set included all SAF participants who comply with the protocol and meet no criteria that could impact the proper evaluation of key objectives of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Late Liver Stage: Pooled Placebo | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
Number analyzed (Participants) | 3 | 3 | 3 | 3
Participants | 3 | 0 | 0 | 0

3. Primary Outcome: Early Liver Stage: Time to First Positive Parasitemia Based on Quantitative Polymerase Chain Reaction (qPCR)
Description: Time to first positive parasitemia was defined as the time (i.e., number of days) from the PfSPZ DVI (i.e., date of DVI PfSPZ) to the first qPCR outcome greater than or equal to (>=) 100 asexual parasites per milliliter (mL) of blood.
Time Frame: Early Liver Stage: From Day 1 up to Day 28
Population: PP analysis set included all SAF participants who comply with the protocol and meet no criteria that could impact the proper evaluation of key objectives of the study. Here, "Overall Number of Participants Analyzed" signifies those participants who had positive parasitemia.
Measure: Median (Full Range); unit: Days
Arm/Group | Early Liver Stage: Pooled Placebo | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717
Number analyzed (Participants) | 6 | 3 | 2 | 1 | 0 | 0
Days | 10.0 [9 to 12] | 15.0 [15 to 18] | 22.0 [20 to 24] | 24.0 [24 to 24] |  |

4. Primary Outcome: Late Liver Stage: Time to First Positive Parasitemia Based on Quantitative Polymerase Chain Reaction (qPCR)
Description: as for outcome 3
Time Frame: Late Liver Stage: From Day 5 up to Day 32
Population: as for outcome 3
Measure: Median (Full Range); unit: Days
Arm/Group | Late Liver Stage: Pooled Placebo | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
Number analyzed (Participants) | 3 | 0 | 0 | 0
Days | 10.0 [9 to 11] |  |  |

5. Primary Outcome: Early Liver Stage: Number of Participants With Documented Blood Stage Parasite Growth
Description: Documented blood stage parasite growth was defined as an increase of qPCR measured asexual parasites per mL compared to the first parasitemia measurement, within 28 days of PfSPZ DVI.
Time Frame: Early Liver Stage: From Day 1 up to Day 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Early Liver Stage: Pooled Placebo | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717
Number analyzed (Participants) | 6 | 3 | 6 | 6 | 3 | 3
Participants | 5 | 2 | 2 | 1 | 0 | 0

6. Primary Outcome: Late Liver Stage: Number of Participants With Documented Blood Stage Parasite Growth
Description: as for outcome 5
Time Frame: Late Liver Stage: From Day 5 up to Day 32
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Late Liver Stage: Pooled Placebo | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
Number analyzed (Participants) | 3 | 3 | 3 | 3
Participants | 3 | 0 | 0 | 0

7. Primary Outcome: Early Liver Stage: Clinical Symptoms of Malaria Assessed Using Malaria Clinical Score
Description: The malaria clinical score consisted of 14 signs/symptoms frequently associated with malaria and graded using a 4-point scale (absent: 0; mild: 1; moderate: 2; severe: 3) and summed to generate a total malaria clinical score (maximum score possible is 42): headache, myalgia (muscle ache), arthralgia (joint ache), fatigue/lethargy, malaise (general discomfort/uneasiness), chills/shivering/rigors, sweating/hot spells, anorexia, nausea, vomiting, abdominal discomfort, fever, tachycardia and hypotension. The minimum score was 0 (no symptoms) and the maximum score was 42 (maximum symptoms). Total scores are reported here.
Time Frame: Early Liver Stage: At Day 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 22, 24, 26 and 28
Population: PP analysis set included all SAF participants who comply with the protocol and meet no criteria that could impact the proper evaluation of key objectives of the study. Here, "Number analyzed" signifies those participants who were evaluable for this outcome at specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a Scale
Arm/Group | Early Liver Stage: Pooled Placebo | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717
Number analyzed (Participants) | 6 | 3 | 6 | 6 | 3 | 3
score on a Scale
  At Day 6 | 0.0 (0.00) | 0.3 (0.58) | 0.2 (0.41) | 0.0 (0.00) | 0.0 (0.00) | 0.1 (0.30)
  At Day 7 | 0.3 (0.52) | 0.3 (0.58) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  At Day 8 | 0.2 (0.41) | 0.3 (0.58) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  At Day 9 | 0.2 (0.41) | 0.3 (0.58) | 0.2 (0.41) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  At Day 10 | 0.3 (0.52) | 0.3 (0.58) | 0.0 (0.00) | 0.3 (0.52) | 0.0 (0.00) | 0.0 (0.00)
  At Day 11 | 0.2 (0.41) | 0.0 (0.00) | 0.0 (0.00) | 0.2 (0.41) | 0.0 (0.00) | 0.0 (0.00)
  At Day 12 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.2 (0.41) | 0.0 (0.00) | 0.0 (0.00)
  At Day 13 | 1.7 (1.86) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  At Day 14 | 4.5 (3.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  At Day 15 | 1.5 (2.07) | 0.0 (0.00) | 0.2 (0.41) | 0.2 (0.41) | 0.0 (0.00) | 0.0 (0.00)
  At Day 16 | 2.0 (1.41) | 0.3 (0.58) | 0.3 (0.52) | 0.2 (0.41) | 0.0 (0.00) | 0.0 (0.00)
  At Day 17 | 0.5 (0.71) | 2.0 (3.46) | 0.3 (0.52) | 0.2 (0.41) | 0.0 (0.00) | 0.0 (0.00)
  At Day 18 | 1.0 (1.41) | 2.3 (4.04) | 0.3 (0.52) | 0.2 (0.41) | 0.3 (0.58) | 0.3 (0.58)
  At Day 19: number analyzed (Participants) | 0 | 3 | 6 | 6 | 3 | 3
  At Day 19 |  | 0.7 (1.15) | 0.3 (0.52) | 0.0 (0.00) | 0.3 (0.58) | 0.0 (0.00)
  At Day 20: number analyzed (Participants) | 0 | 3 | 6 | 6 | 3 | 3
  At Day 20 |  | 1.0 (1.73) | 0.0 (0.00) | 0.0 (0.00) | 0.3 (0.58) | 0.0 (0.00)
  At Day 22 | 0.0 (0.00) | 0.7 (1.15) | 0.0 (0.00) | 0.2 (0.41) | 0.0 (0.00) | 0.0 (0.00)
  At Day 24: number analyzed (Participants) | 0 | 0 | 6 | 6 | 3 | 3
  At Day 24 |  |  | 0.0 (0.00) | 0.2 (0.41) | 0.0 (0.00) | 0.0 (0.00)
  At Day 26 | 0.0 (0.00) | 0.0 (0.00) | 0.2 (0.41) | 0.2 (0.41) | 0.0 (0.00) | 0.3 (0.58)
  At Day 28 | 0.0 (0.0) | 0.0 (0.00) | 0.2 (0.41) | 0.2 (0.41) | 0.3 (0.58) | 0.0 (0.00)

8. Primary Outcome: Late Liver Stage: Clinical Symptoms of Malaria Assessed Using Malaria Clinical Score
Description: as for outcome 7
Time Frame: Late Liver Stage: At Day 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 26, 28, 30 and 32
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Late Liver Stage: Pooled Placebo | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
Number analyzed (Participants) | 3 | 3 | 3 | 3
Score on a Scale
  At Day 6 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  At Day 7 | 0.0 (0.00) | 0.3 (0.58) | 0.0 (0.00) | 0.0 (0.00)
  At Day 8 | 0.0 (0.00) | 0.0 (0.00) | 0.3 (0.58) | 0.0 (0.00)
  At Day 9 | 0.3 (0.58) | 0.0 (0.00) | 0.3 (0.58) | 0.0 (0.00)
  At Day 10 | 0.3 (0.58) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  At Day 11 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  At Day 12 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  At Day 13 | 0.0 (0.00) | 0.3 (0.58) | 0.0 (0.00) | 0.0 (0.00)
  At Day 14 | 0.0 (0.00) | 0.0 (0.00) | 0.3 (0.58) | 0.0 (0.00)
  At Day 15 | 1.5 (2.12) | 0.0 (0.00) | 0.3 (0.58) | 0.3 (0.58)
  At Day 16 | 1.5 (2.12) | 0.3 (0.58) | 0.0 (0.00) | 0.0 (0.00)
  At Day 17: number analyzed (Participants) | 1 | 3 | 3 | 3
  At Day 17 | 1.0 | 0.0 (0.00) | 0.3 (0.58) | 0.7 (1.15)
  At Day 18: number analyzed (Participants) | 0 | 3 | 3 | 3
  At Day 18 |  | 0.3 (0.58) | 0.3 (0.58) | 0.0 (0.00)
  At Day 19 | 0.0 (0.00) | 0.0 (0.00) | 0.3 (0.58) | 0.0 (0.00)
  At Day 20: number analyzed (Participants) | 0 | 3 | 3 | 3
  At Day 20 |  | 0.0 (0.00) | 0.3 (0.58) | 0.0 (0.00)
  At Day 21: number analyzed (Participants) | 0 | 3 | 3 | 3
  At Day 21 |  | 0.3 (0.58) | 0.3 (0.58) | 0.3 (0.58)
  At Day 22: number analyzed (Participants) | 0 | 3 | 3 | 3
  At Day 22 |  | 0.0 (0.00) | 0.3 (0.58) | 0.3 (0.58)
  At Day 23: number analyzed (Participants) | 0 | 3 | 3 | 3
  At Day 23 |  | 0.0 (0.00) | 0.0 (0.00) | 0.3 (0.58)
  At Day 24: number analyzed (Participants) | 0 | 3 | 3 | 3
  At Day 24 |  | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  At Day 26 | 0.3 (0.58) | 0.3 (0.58) | 0.0 (0.00) | 0.0 (0.00)
  At Day 28: number analyzed (Participants) | 0 | 3 | 3 | 3
  At Day 28 |  | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  At Day 30 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.00 (0.00)
  At Day 32 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious TEAEs and Treatment-related TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered with study drug which does not necessarily had a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAE was defined as AEs starting or worsening after the first intake of the study drug. TEAEs included both serious TEAEs and non-serious TEAEs. Treatment-related TEAEs: reasonably related to study intervention.
Time Frame: Early Liver Stage: From Day 1 up to Day 33; Late Liver Stage: From Day 1 up to Day 36
Population: SAF included all ITT participants, who have been inoculated using a Direct Intravenous Inoculation (DVI) of PfSPZ and who were administered one dose of study intervention (M5717 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Early Liver Stage: Pooled Placebo | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717 | Late Liver Stage: Pooled Placebo | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
Number analyzed (Participants) | 6 | 3 | 6 | 6 | 3 | 3 | 3 | 3 | 3 | 3
Participants
  Participants with TEAEs | 5 | 3 | 6 | 6 | 3 | 3 | 3 | 3 | 2 | 2
  Participants with Serious TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants with Treatment-related TEAEs | 2 | 0 | 2 | 2 | 1 | 3 | 0 | 1 | 0 | 0

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Based on Severity
Description: Severity of adverse events (AE) were assessed by the investigator per the Qualitative Toxicity Scale. Grade 1= Mild, Grade 2=Moderate, Grade 3=Severe. The number of participants that experienced at least one solicited local TEAE were summarized by grade. The term TEAE is defined as AEs starting or worsening after the first intake of the study drug. TEAEs include both Serious TEAEs and non-serious TEAEs. Number of participants with Grade=1, Grade=2 and 3 were reported.
Time Frame: Early Liver Stage: From Day 1 up to Day 33; Late Liver Stage: From Day 1 up to Day 36
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Early Liver Stage: Pooled Placebo | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717 | Late Liver Stage: Pooled Placebo | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
Number analyzed (Participants) | 6 | 3 | 6 | 6 | 3 | 3 | 3 | 3 | 3 | 3
Participants
  Grade 1 (Mild) | 5 | 3 | 6 | 6 | 3 | 3 | 3 | 3 | 2 | 2
  Grade 2 (Moderate) | 3 | 2 | 2 | 1 | 0 | 1 | 2 | 0 | 0 | 0
  Grade 3 (Severe) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Laboratory Values
Description: Laboratory assessments included hematology, biochemistry, urinalysis, and coagulation. Number of participants with clinically significant changes from baseline in laboratory values which were deemed clinically significant by the investigator were reported.
Time Frame: Early Liver Stage: From Day 1 up to Day 33; Late Liver Stage: From Day 1 up to Day 36
Population: SAF included all ITT participants, who have been inoculated using a DVI of PfSPZ and who were administered one dose of study intervention (M5717 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Early Liver Stage: Pooled Placebo | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717 | Late Liver Stage: Pooled Placebo | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
Number analyzed (Participants) | 6 | 3 | 6 | 6 | 3 | 3 | 3 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs included oral body temperature, height, weight, systolic blood pressure, diastolic blood pressure, and pulse rate. Number of participants with clinically significant changes from baseline in Vital signs which were deemed clinically significant by the investigator were reported.
Time Frame: Early Liver Stage: From Day 1 up to Day 33; Late Liver Stage: From Day 1 up to Day 36
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Early Liver Stage: Pooled Placebo | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717 | Late Liver Stage: Pooled Placebo | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
Number analyzed (Participants) | 6 | 3 | 6 | 6 | 3 | 3 | 3 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in 12-lead Electrocardiogram (ECG) Findings
Description: Single 12-lead ECG was obtained as outlined using an ECG machine that automatically calculates the heart rate and measures PR, QRS, and QT intervals. Number of participants with clinically significant changes from baseline in ECG which were deemed clinically significant by the investigator were reported.
Time Frame: Early Liver Stage: From Day 1 up to Day 33; Late Liver Stage: From Day 1 up to Day 36
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Early Liver Stage: Pooled Placebo | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717 | Late Liver Stage: Pooled Placebo | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
Number analyzed (Participants) | 6 | 3 | 6 | 6 | 3 | 3 | 3 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Area Under the Blood Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of M5717
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUC extra represents an extrapolated value obtained by Clast/ λz, where Clast is the calculated blood concentration at the last sampling time point at which the measured blood concentration is at or above the Lower Limit of quantification (LLQ) and λz is the apparent terminal rate constant determined by log-linear regression analysis of the measured blood concentrations of the terminal log-linear phase.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 6, 12, 24, 120, 168, 192, 600, and 768 hours post-dose
Population: PK analysis set included all participants, who received 1 dose of M5717, had no clinically important protocol deviations/important events affecting PK, & provide at least 1 measurable post-dose concentration. Data was not available for 'Early liver stage: 30 mg M5717' arm as no participants were considered evaluable because of limited number of samples collected to characterize the elimination rate constant (lambda z) needed for calculation of AUC0-inf.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter(hour*ng/mL)
Arm/Group | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717 | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
Number analyzed (Participants) | 0 | 6 | 6 | 3 | 3 | 3 | 3 | 3
hour*nanogram per milliliter(hour*ng/mL) |  | 1280 (31.81) | 1990 (25.24) | 1890 (12.52) | 9840 (37.44) | 1100 (71.03) | 2330 (4.70) | 4830 (53.73)

15. Secondary Outcome: Area Under the Blood Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC 0-tlast) of M5717
Description: Area under the blood concentration vs time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLQ). AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 6, 12, 24, 120, 168, 192, 600, and 768 hours post-dose
Population: Pharmacokinetic analysis set included all participants, who received one dose of M5717, have no clinically important protocol deviations or important events affecting PK, and provide at least one measurable post-dose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717 | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
Number analyzed (Participants) | 3 | 6 | 6 | 3 | 3 | 3 | 3 | 3
hour*ng/mL | 21.9 (1160.32) | 852 (36.35) | 1270 (14.08) | 1470 (4.65) | 7330 (42.80) | 657 (67.17) | 1810 (8.09) | 3820 (70.38)

16. Secondary Outcome: Area Under the Blood Concentration-Time Curve From Time Zero to 24 Hours Post-dose (AUC 0-24) of M5717
Description: AUC from time zero to 24 hours post dose, calculated using the mixed log linear trapezoidal rule (linear up, log down) using the nominal dosing interval.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 6, 12 and 24 hours post-dose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717 | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
Number analyzed (Participants) | 3 | 6 | 6 | 3 | 3 | 3 | 3 | 3
h*ng/mL | 25.8 (639.59) | 198 (40.21) | 280 (18.23) | 290 (39.80) | 975 (33.02) | 160 (44.63) | 445 (8.60) | 1020 (45.85)

17. Secondary Outcome: Area Under the Blood Concentration-Time Curve From Time Zero to 168 Hours Post-dose (AUC 0-168) of M5717
Description: AUC from time zero to 168 hours post dose. Calculated using the mixed log linear trapezoidal rule (linear up, log down) using the nominal dosing interval.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 6, 12, 24, 120 and 168 hours post-dose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717 | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
Number analyzed (Participants) | 3 | 6 | 6 | 3 | 3 | 3 | 3 | 3
h*ng/mL | 50.4 (2325.31) | 805 (35.22) | 1190 (14.35) | 1390 (5.34) | 3680 (29.33) | 692 (53.24) | 1710 (8.67) | 3190 (43.40)

18. Secondary Outcome: Maximum Observed Blood Concentration (Cmax) of M5717
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 6, 12, 24, 120, 168, 192, 600, and 768 hours post-dose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717 | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
Number analyzed (Participants) | 3 | 6 | 6 | 3 | 3 | 3 | 3 | 3
nanogram per milliliter (ng/mL) | 3.56 (39.90) | 11.7 (36.93) | 16.6 (33.70) | 17.2 (44.12) | 57.2 (38.08) | 9.38 (82.50) | 27.6 (22.19) | 64.4 (46.26)

19. Secondary Outcome: Blood Concentration at 24 Hours (C24) of M5717
Description: Blood samples for PK analysis of C24 of M5717 was reported.
Time Frame: At 24 hours post-dose
Population: Pharmacokinetic analysis set included all participants, who received one dose of M5717, have no clinically important protocol deviations or important events affecting PK, and provide at least one measurable post-dose concentration. Here, "Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717 | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
Number analyzed (Participants) | 2 | 6 | 6 | 3 | 3 | 3 | 3 | 3
ng/mL | NA (NA) — Based on pre-specified criteria Geometric Mean and Geometric Coefficient of Variation were not calculated if fewer than 3 participants have reportable parameter values. | 6.77 (45.35) | 9.42 (28.12) | 11.3 (31.42) | 30.6 (24.91) | 6.06 (37.89) | 14.9 (14.56) | 26.7 (37.88)

20. Secondary Outcome: Blood Concentration at 168 Hours (C168) of M5717
Description: C168 is the calculated blood concentration at 168 hours post-dose at which the measured blood concentration is at or above the Lower Limit of quantification (LLQ).
Time Frame: At 168 hours post-dose
Population: PK analysis set included all participants, who received one dose of M5717, have no clinically important protocol deviations or important events affecting PK, & provide at least one measurable post-dose concentration. "Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717 | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
Number analyzed (Participants) | 3 | 6 | 6 | 3 | 3 | 1 | 3 | 3
ng/mL | NA (NA) — Data was not calculable as the concentration was at below the lower limit of quantification. | 2.89 (38.61) | 4.31 (13.43) | 4.16 (24.60) | 11.4 (40.64) | NA (NA) — Based on pre-specified criteria Geometric Mean and Geometric Coefficient of Variation were not calculated if fewer than 3 participants have reportable parameter values. | 4.88 (2.50) | 8.30 (45.60)

21. Secondary Outcome: Time to Reach Maximum Blood Concentration (Tmax) of M5717
Description: Time to reach the maximum blood concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 6, 12, 24, 120, 168, 192, 600, and 768 hours post-dose
Population: as for outcome 15
Measure: Median (Full Range); unit: Hours
Arm/Group | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717 | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
Number analyzed (Participants) | 3 | 6 | 6 | 3 | 3 | 3 | 3 | 3
Hours | 6.00 [0.500 to 12.0] | 1.00 [0.500 to 12.0] | 3.25 [0.500 to 12.0] | 6.00 [0.500 to 12.0] | 1.00 [0.500 to 6.00] | 1.00 [0.500 to 1.00] | 2.00 [1.00 to 2.02] | 2.00 [2.00 to 2.00]

22. Secondary Outcome: Apparent Terminal Half-life (t1/2) of M5717
Description: Terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by lambda z.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 6, 12, 24, 120, 168, 192, 600, and 768 hours post-dose
Population: PK analysis set included all participants, who received 1 dose of M5717, had no clinically important protocol deviations/important events affecting PK, & provide at least 1 measurable post-dose concentration. Data was not available for 'Early liver stage: 30 mg M5717' arm as no participants were considered evaluable because of limited number of samples collected to characterize the elimination rate constant (lambda z) needed for calculation of t1/2.
Measure: Median (Full Range); unit: Hours
Arm/Group | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717 | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
Number analyzed (Participants) | 0 | 6 | 6 | 3 | 3 | 3 | 3 | 3
Hours |  | 121 [82.3 to 143] | 121 [97.2 to 221] | 66.9 [66.6 to 108] | 494 [212 to 531] | 94.1 [74.2 to 156] | 95.4 [76.0 to 95.5] | 136 [101 to 183]

23. Secondary Outcome: Elimination Rate Constant (Lambda z) of M5717
Description: Elimination rate constant determined from the terminal slope of the log-transformed concentration curve using linear regression on terminal data points of the curve.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 6, 12, 24, 120, 168, 192, 600, and 768 hours post-dose
Population: PK analysis set included all participants, who received 1 dose of M5717, had no clinically important protocol deviations/important events affecting PK, & provide at least 1 measurable post-dose concentration. Data was not available for 'Early liver stage: 30 mg M5717' arm as no participants were considered evaluable because of limited number of samples collected to characterize the elimination rate constant (lambda z).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: One per Hours (1/h)
Arm/Group | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717 | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
Number analyzed (Participants) | 0 | 6 | 6 | 3 | 3 | 3 | 3 | 3
One per Hours (1/h) |  | 0.00597 (22.93) | 0.00529 (30.44) | 0.00885 (28.59) | 0.00182 (55.45) | 0.00677 (38.43) | 0.00786 (12.78) | 0.00511 (30.50)

24. Secondary Outcome: Apparent Total Body Clearance From Blood (CL/f) of M5717
Description: Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Apparent body clearance of the drug from blood, CL= Dose/AUC0-inf
Time Frame: Pre-dose, 0.5, 1, 2, 3, 6, 12, 24, 120, 168, 192, 600, and 768 hours post-dose
Population: PK analysis set included all participants, who received 1 dose of M5717, had no clinically important protocol deviations/important events affecting PK, & provide at least 1 measurable post-dose concentration. Data was not available for 'Early liver stage: 30 mg M5717' arm as no participants were considered evaluable because of limited number of samples collected to characterize the elimination rate constant (lambda z) needed for calculation of CL/f.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per Hours (L/h)
Arm/Group | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717 | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
Number analyzed (Participants) | 0 | 6 | 6 | 3 | 3 | 3 | 3 | 3
Liter per Hours (L/h) |  | 46.9 (31.81) | 40.3 (25.24) | 52.9 (12.52) | 20.3 (37.44) | 54.8 (71.03) | 43.0 (4.70) | 41.4 (53.73)

25. Secondary Outcome: Apparent Volume of Distribution (Vz/F) During the Terminal Phase of M5717
Description: The Vz/f was defined as the theoretical volume in which the total amount of required to uniformly distribute to produce the desired plasma concentration. Apparent volume of distribution after oral dose (Vz/F) was influenced by the fraction absorbed. The Vz/f was calculated by dividing the dose with area under the concentration time curve from time zero to infinity multiplied with terminal elimination rate constant Lambda(z). Vz/f=Dose/AUC(0-inf) multiply Lambda(z).
Time Frame: Pre-dose, 0.5, 1, 2, 3, 6, 12, 24, 120, 168, 192, 600, and 768 hours post-dose
Population: PK analysis set included all participants, who received 1 dose of M5717, had no clinically important protocol deviations/important events affecting PK, & provide at least 1 measurable post-dose concentration. Data was not available for 'Early liver stage: 30 mg M5717' arm as no participants were considered evaluable because of limited number of samples collected to characterize the elimination rate constant (lambda z) needed for calculation of Vz/F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717 | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
Number analyzed (Participants) | 0 | 6 | 6 | 3 | 3 | 3 | 3 | 3
Liter |  | 7850 (42.71) | 7600 (10.87) | 5980 (15.57) | 11200 (60.47) | 8130 (35.29) | 5490 (15.71) | 27.59 (8340)

26. Primary Outcome: Dose Exposure Response Relationship of M5717 Assessed by Logistic Regression Model
Description: Exposure efficacy relationship was analyzed using logistic regression model. Different exposure matrices (AUC0-24, AUC0-168, AUC0-inf, C24 and C168) were analyzed using logistic regression model.
Time Frame: From Day 5 up to Day 32
Population: PP analysis set included all SAF participants who comply with protocol and meet no criteria that could impact proper evaluation of key objectives of study. This data was analyzed together jointly across cohorts and hence model parameter were based on complete data set as opposed to cohort by cohort.
Measure: Number; unit: slope
Groups:
- All Participants: AUC0-24; All Participants: AUC0-168; All Participants: AUC0-inf; All Participants: C24; All Participants: C168: Participants received single dose of placebo matched to M5717 or 30 mg or 60 mg or 80 mg or 100 mg or 200 mg of M5717 capsule during early liver stage on Day 1 after 2 hours of PfSPZ IV inoculation administration on Day 1 or received single dose of placebo matched to M5717 or 60 mg or 100 mg or 200 mg of M5717 capsule during the late liver stage on Day 5 after 96 hours of PfSPZ IV inoculation administration on Day 1.
Arm/Group | All Participants: AUC0-24 | All Participants: AUC0-168 | All Participants: AUC0-inf | All Participants: C24 | All Participants: C168
Number analyzed (Participants) | 39 | 39 | 39 | 39 | 39
slope | 1.27 | 1.43 | 1.44 | 0.800 | 2.45
Statistical Analysis 1: Comparison: All Participants: AUC0-24; Test type: Other; p = 0.00284, Regression, Logistic; Odds Ratio (OR) = 3.57, 95% CI 2-sided [1.85 to 10.6]
Statistical Analysis 2: Comparison: All Participants: AUC0-168; Test type: Other; p = 0.00367, Regression, Logistic; Odds Ratio (OR) = 4.19, 95% CI 2-sided [2.00 to 14.8]
Statistical Analysis 3: Comparison: All Participants: AUC0-inf; Test type: Other; p = 0.0137, Regression, Logistic; Odds Ratio (OR) = 4.22, 95% CI 2-sided [1.90 to 23.7]
Statistical Analysis 4: Comparison: All Participants: C24; Test type: Other; p = 0.00349, Regression, Logistic; Odds Ratio (OR) = 2.23, 95% CI 2-sided [1.47 to 4.48]
Statistical Analysis 5: Comparison: All Participants: C168; Test type: Other; p = 0.00594, Regression, Logistic; Odds Ratio (OR) = 11.6, 95% CI 2-sided [3.19 to 129]

ADVERSE EVENTS:
Time Frame: Early Liver Stage: From Day 1 up to Day 33; Late Liver Stage: From Day 1 up to Day 36
Arm/Group | Early Liver Stage: Pooled Placebo | Early Liver Stage: 30 mg M5717 | Early Liver Stage: 60 mg M5717 | Early Liver Stage: 80 mg M5717 | Early Liver Stage: 100 mg M5717 | Early Liver Stage: 200 mg M5717 | Late Liver Stage: Pooled Placebo | Late Liver Stage: 60 mg M5717 | Late Liver Stage: 100 mg M5717 | Late Liver Stage: 200 mg M5717
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/6 | 0/6 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/6 | 0/6 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 5/6 | 3/3 | 6/6 | 6/6 | 3/3 | 3/3 | 3/3 | 3/3 | 2/3 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early Liver Stage: Pooled Placebo (N=6) | Early Liver Stage: 30 mg M5717 (N=3) | Early Liver Stage: 60 mg M5717 (N=6) | Early Liver Stage: 80 mg M5717 (N=6) | Early Liver Stage: 100 mg M5717 (N=3) | Early Liver Stage: 200 mg M5717 (N=3) | Late Liver Stage: Pooled Placebo (N=3) | Late Liver Stage: 60 mg M5717 (N=3) | Late Liver Stage: 100 mg M5717 (N=3) | Late Liver Stage: 200 mg M5717 (N=3)
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 3 | 2 | 2 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 0 | 4 | 1 | 2 | 1 | 3 | 2 | 1 | 2
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 4 | 2 | 3 | 3 | 2 | 2 | 2 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 4 | 3 | 1 | 1 | 0 | 2 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 2 | 1 | 0 | 1 | 0 | 1 | 3 | 0 | 1
Feeling cold (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Tenderness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT04250363/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT04250363/SAP_001.pdf